CLINICAL TRIAL: NCT03782311
Title: The Relationship Between Oral Hygiene Related Self-efficacy, General Self-efficacy and Daily Plaque Control
Brief Title: Oral Hygiene Related Self-efficacy, General Self-efficacy and Daily Plaque Control
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gul Atilla, Clinical Professor, Ege University
Other Study IDs: c37taicm
Record Dates: First submitted 2018-12-15; First posted 2018-12-20 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Dental Plaque
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 2 groups: OHSE-high and OHSE-low: OHSE-high: Group with ≥ 50 OHSE scores received motivation and oral hygiene instructions .
  OHSE-low: Group with < 30 OHSE scores received motivation and oral hygiene instructions .
  Interventions: Behavioral: motivation and and oral hygiene instructions

INTERVENTIONS:
Behavioral: motivation and and oral hygiene instructions — Motivation and oral hygiene instructions were received OHSE-high and OHSE-low groups. After showing the modified-Bass tooth brushing technique and interdental cleaning on the model, patients were followed up while brushing and flossing their teeth to correct misapplications. It was advised to brush teeth twice a day and use the interdental cleaning devices once a day.

SUMMARY:
The objectives are a) to determine the scores of general self-efficacy (GSE) and oral hygiene related self-efficacy (OHSE) b) to evaluate the relations between the scores of GSE and OHSE c) to examine the changes in OHSE scores and the relationship between OHSE and PI scores after motivation and oral hygiene instructions. OHSE scores could be an indicator in predicting daily plaque control of patients. Also, it may be needed to show greater interest about motivation and oral hygiene instructions especially for smokers and OHSE-low group patients.

DETAILED DESCRIPTION:
All study patients (n=210) between the ages of 35 to 60 with inflammatory periodontal diseases filled out questionnaires regarding GSE and OHSE. Subgroups including OHSE-low (n=26) and OHSE-high (n=26) groups were selected after performing "cut off" on OHSE scores of all study patients. In both subgroups, plaque index (PI) values were determined, and motivation and oral hygiene instructions were performed at baseline. PI measurements and OHSE questionnaire were repeated at 1 and 3 months.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria were being able to brushing and interdental cleaning physically and mentally, between the ages of 35 and 60, graduated from high school or university, having at least 12 teeth, no periodontal treatment in the last 6 months, no periodontal surgery in the last 2 years.

Exclusion Criteria:

Patients with one or more of the following criteria were excluded from the study: patients having hepatitis or HIV infectious disease, pregnant and lactating females, patients taking drugs that may cause gingival bleeding and gingival enlargement, and bleeding problems (thrombocytopenia, hemophilia A-B, iron deficiency anemia etc.).

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Gingivitis and periodontitis patients
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
oral hygiene related self-efficacy (OHSE) score (min:19, max:76, higher values represent a better ), summed | baseline
  Woelber et al. in 2015
"change" is being assessed. oral hygiene related self-efficacy (OHSE) score (min:19, max:76, higher values represent a better), summed | 1 mouth
  Woelber et al. in 2015
"change" is being assessed. oral hygiene related self-efficacy (OHSE) score (min:19, max:76, higher values represent a better ), summed | 3 mouth
  Woelber et al. in 2015
plaque index (min:0, max:5, lower values represent a better), averaged | baseline
  Quigley & Hein (1962) Plaque Index
"change" is being assessed. plaque index (min:0, max:5, lower values represent a better), averaged | 1 month
  Quigley & Hein (1962) Plaque Index
"change" is being assessed. plaque index (min:0, max:5, lower values represent a better), averaged | 3 month
  Quigley & Hein (1962) Plaque Index

SECONDARY OUTCOMES:
General Self Efficacy (GSE) score (min:10, max: 40), summed | baseline
  Schwarzer & Jerusalem, 1995
Demographic variables | baseline
  age, gender, smoking, number of teeth, education, income

CONTACTS AND LOCATIONS:
Overall Officials: Gul Atilla, Principal Investigator — clinical professor